CLINICAL TRIAL: NCT00621751
Title: Carbamazepine for the Treatment of Chronic Post-Traumatic Brain Injury Irritability and Aggression: A 42-Day, Single-Site, Forced-Titration, Parallel Group, Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Carbamazepine for the Treatment of Chronic Post-Traumatic Brain Injury Irritability and Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-07-02A; H133A20016 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-08

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injury; Irritability; Aggression
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Aggression | interventions — Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbamazepine (Experimental): Carbamazepine 800 mg daily
  Interventions: Drug: Carbamazepine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbamazepine — 800 mg daily
  Other Names: Tegretol
  Arms: Carbamazepine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if carbamazepine reduces irritability and aggression among individuals with traumatic brain injury

DETAILED DESCRIPTION:
To achieve the enrollment of 66 needed, over enrollment of 70 subjects with 70 corresponding subject informants will be recruited at Carolinas Rehabilitation. Subjects will be recruited from the clinic at Carolinas Rehabilitation. Subjects will also be referred by psychiatrists at North Carolina Neuropsychiatry.

Subjects who consent and qualify will be randomized in a 1:1 ratio to Tegretol® or placebo. Stratification to randomization group will occur based on the presence of depression defined by a Beck Depression Inventory-II score ≥ 13. Subjects randomized to active drug will be titrated up in dose, as tolerated, over a period of 3 weeks. Starting dose is 200mg twice daily to 200mg three times daily to 200mg, 2 tabs, twice daily. There will be 3 clinic visits. Visits will occur at baseline for consenting and screening, day 28, and day 42. Follow up phone calls will occur each week that the subject is not seen in the clinic until the end of the study. Follow up phone calls will assess for study medication compliance, adverse events and concomitant medication changes. Day 42 ends the period of the Randomized Clinical Trial phase of the study and the subjects will begin the 1 week of taper of Tegretol® at 400mg daily and then stop drug. A safety phone call will be made at day 49.

The following questionnaires will be used as measures of irritability for the subject and the informant: Neuropsychiatric Inventory (NPI), and Global Impression of Change. The Beck Depression Inventory will be administered to the participant only at baseline for purposes of stratification of the randomization on depression. The Clinician Investigator will complete the Clinician Global Impressions scale at Visits 2 and 3.

History and Physical Exam, hematology, chemistry, including renal and liver function studies will be obtained for safety and tolerability. Serum pregnancy tests will be drawn at screening for females of childbearing potential. Carbamazepine levels will be drawn at visits 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Closed head injury (defined as impaired brain function resulting from externally inflicted trauma without penetrating injury) at least 6 months prior to enrollment
* Age at time of enrollment: 16 to 75 years
* Voluntary informed consent of patient and informant
* Subject and informant willing to comply with the protocol
* Informant-rated NPI Irritability Domain score 6 or greater to include only moderate-severe irritability
* Medically and neurologically stable during the month prior to enrollment If taking antidepressant, anxiolytic, hypnotic, or stimulant medications, no change anticipated in these medications during the month prior to enrollment No change in therapies or medications planned during the 42-day participation No surgeries planned during the 42-day participation Vision, hearing, speech, motor function, and comprehension sufficient for compliance with all testing procedures and assessments
* Informant (e.g. family member or close friend) with daily interaction in order to observe occurrences of irritability

Exclusion Criteria:

* Potential subject without a reliable informant
* Penetrating head injury
* Injury < 6 months prior to enrollment
* Ingestion of carbamazepine during the month prior to enrollment
* Inability to interact sufficiently for communication with caregiver
* Acute and rehabilitation records unavailable or incomplete
* Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of schizophrenia or psychosis
* Diagnosis of progressive or additional neurologic disease
* Clinical signs of active infection
* Creatinine clearance <60 mL/min
* Liver function tests > 2x normal values
* Pregnancy; lactating females; sexually active females who do not agree to use birth control
* Hormonal birth control as only means of birth control if sexually active and of child bearing age potential due to carbamazepine effect of lowering hormone levels, and potentially effectiveness
* Concurrent use of the following medicines due to potential for drug interaction: macrolides, rifabutin, doxycycline, nicoumalone, warfarin, fluoxetine, fluvoxamine, viloxazine, nefazodone, tricyclic and tetracyclic antidepressants, clobazam, clonazepam, lamotrigine, phenytoin, sodium valproate, tigabine and topiramate, phenobarbitone, primidone, chloroquine and mefloquine, antipsychotics, indinavir, nelfinavir, saquinavir, ritonavir, diltiazem, verapamil, felodipine, isradipine, nicardipine, nifedipine, cimetidine, cyclosporins, corticosteroids, gestrinone and toremifene, danazol, tibolone
* Suicidal ideation
* Concurrent use of Monoamine Oxidase Inhibitors or ingestion of within 2 weeks before starting study
* Hypersensitivity/allergy to carbamazepine, any of the ingredients in carbamazepine, or any structurally related drugs (e.g. the tricyclic antidepressants)
* History of liver failure or hepatitis
* History of renal failure
* History atrio-ventricular conduction abnormalities unless paced
* History of bone marrow depression
* History of porphyria
* Asian heritage

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-02; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flora M Hammond, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Azouvi P, Jokic C, Attal N, Denys P, Markabi S, Bussel B. Carbamazepine in agitation and aggressive behaviour following severe closed-head injury: results of an open trial. Brain Inj. 1999 Oct;13(10):797-804. doi: 10.1080/026990599121188. PMID 10576463
- [Background] Chatham-Showalter PE. Carbamazepine for combativeness in acute traumatic brain injury. J Neuropsychiatry Clin Neurosci. 1996 Winter;8(1):96-9. doi: 10.1176/jnp.8.1.96. PMID 8845710
- [Background] Lewin J, Sumners D. Successful treatment of episodic dyscontrol with carbamazepine. Br J Psychiatry. 1992 Aug;161:261-2. doi: 10.1192/bjp.161.2.261. PMID 1521112
- [Background] Wroblewski BA, Joseph AB, Kupfer J, Kalliel K. Effectiveness of valproic acid on destructive and aggressive behaviours in patients with acquired brain injury. Brain Inj. 1997 Jan;11(1):37-47. doi: 10.1080/026990597123791. PMID 9012550
- See also: Carolinas Rehabilitation — http://www.carolinasrehabilitation.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbamazepine | Placebo
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbamazepine | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.9) | 40.5 (13.7) | 40.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 35 | 33 | 68
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 28 | 24 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychiatric Inventory Irritability-Aggression Domains Composite Measure -- Observer
Description: Neuropsychiatry Inventory-Irritability (NPI-I) & Aggression domains (NPI-A): NPI is a 40-item assessment of 12 behavioral domains (NPI-I & NPI-A domains used in this study). The most problematic aspect of each domain is graded for severity (1=mild, to 3=severe) and frequency (1-4 with 4 representing highest frequency); the domain scores (0-12) are the product of severity and frequency. To best reflect treatment target intent and meet parametric statistical method criteria, the primary outcome was a composite measure of observer-rated NPI-I & -A domains transformed to a Rasch logit scale running from 0 (best) to 100 (worse) units (i.e., observer-rated NPI-I/A Rasch construct scores). Mean day-42 observer-rated NPI-I/A Rasch construct scores were compared between placebo vs. carbamazepine using ANCOVA with baseline score as covariate.
Time Frame: 42 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 35 | 34
score on a scale | 37.7 (1.4) | 36.7 (1.5)
Statistical Analysis 1: Comparison: Carbamazepine vs Placebo; The primary outcome was a composite measure of observer-rated NPI-I & NPI-A domains transformed to a Rasch logit scale ranging 0 (best) to 100 (worse) units (i.e., observer-rated NPI-I/A Rasch construct scores). Mean day-42 observer-rated NPI-I/A Rasch construct scores were compared between the placebo vs. carbamazepine groups using ANCOVA with baseline score as covariate; Test type: Other; p = 0.60, ANCOVA — CBZ (up to 800 mg daily) vs placebo significantly improves behavior (Rasch NPI irritability & aggression rated by observer) baseline to day-42 among individuals >6 months post-traumatic brain injury and moderate-severe irritability; Median Difference (Final Values) = 36.7

2. Secondary Outcome: Proportion of Participants With Minimal Clinically Important Difference -- Observer Rating
Description: Proportion of participants with Minimal Clinically Important Difference (MCID) on Neuropsychiatric Inventory Irritability-Aggression Composite Measure completed by Observer. Specifically, the proportion of participants that experienced a decrease of > 1 (MCID) in the NPI-I/A Rasch construct score (i.e., participants that are considered to have meaningful reduction in irritability/aggression) from baseline to day-42 between the groups using a chi-square test. MCID was defined as 0.5 times the standard deviation of baseline scores.
Time Frame: 42-day
Measure: Count of Participants; unit: Participants
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 35 | 34
Participants | 20 | 26
Statistical Analysis 1: Comparison: Carbamazepine vs Placebo; Test type: Other — A prespecified secondary analysis compared proportions of participants that experienced a decrease of > 1 MCID in the NPI-I/A Rasch construct score (i.e., participants that are considered to have meaningful reduction in irritability/aggression) from baseline to day-42 between the groups using a chi-square test. MCID was defined as 0.5 times the standard deviation of baseline scores; p < .05, ANCOVA

3. Secondary Outcome: Global Impression of Change -- Observer
Description: Global Impression of Change (GIC) is a 5-item Likert Scale rated participants and observer impression of change in the person with TBI. Responses range 1 = much improved to 5 = much worse.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 35 | 34
units on a scale | 3.3 (1.4) | 3.1 (0.9)

4. Secondary Outcome: Neuropsychiatric Inventory Irritability-Aggression Domains Composite Measure Completed by Participant [Time Frame: 42 Days]
Description: Neuropsychiatry Inventory-Irritability (NPI-I) & Aggression domains (NPI-A): NPI is a 40-item assessment of 12 behavioral domains (NPI-I & NPI-A domains used in this study). The most problematic aspect of each domain is graded for severity (1=mild, to 3=severe) and frequency (1-4 with 4 representing highest frequency); the domain scores (0-12) are the product of severity and frequency. To best reflect treatment target intent and meet parametric statistical method criteria, a composite measure of participant-rated NPI-I & -A domains transformed to a Rasch logit scale running from 0 (best) to 100 (worse) units (i.e., participant-rated NPI-I/A Rasch construct scores). Mean day-42 participant-rated NPI-I/A Rasch construct scores were compared between placebo vs. CBZ using ANCOVA with baseline score as covariate.
Time Frame: Day 42
Population: There were fewer participants scores than observers scores.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 32 | 30
score on a scale | 37.5 (1.4) | 36.4 (1.4)

5. Secondary Outcome: Proportion of Participants With Minimal Clinically Important Difference (MCID) -- Participant
Description: Proportion of participants with Minimal Clinically Important Difference (MCID) on Neuropsychiatric Inventory Irritability-Aggression Composite Measure completed by Participant. Specifically, the proportion of participants that experienced a decrease of > 1 (MCID) in the NPI-I/A Rasch construct score (i.e., participants that are considered to have meaningful reduction in irritability/aggression) from baseline to day-42 between the groups using a chi-square test. MCID was defined as 0.5 times the standard deviation of baseline scores.
Time Frame: Day-42
Measure: Count of Participants; unit: Participants
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 32 | 30
Participants | 21 | 16

6. Secondary Outcome: Clinicians Global Impression of Change
Description: Study physician's impression of change since study onset. Clinicians Global Impressions of Change (CGI) is a sensitive, standardized tool to assess psychopharmacologic treatment response completed by the study physician. The Global Improvement (GI) CGI subscale documented the clinician's impression of change. The GI uses a 7-point scale to assess beneficial and negative effects. Low GI values (1 -3) indicate improvement; higher values (4-7) represent worsening.
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 35 | 34
units on a scale | 3.1 (1.3) | 2.9 (1.1)

7. Secondary Outcome: Global Impression of Change -- Participant
Description: as for outcome 3
Time Frame: Day-42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carbamazepine | Placebo
Number analyzed (Participants) | 32 | 30
score on a scale | 3.1 (1.3) | 3.1 (0.9)

ADVERSE EVENTS:
Time Frame: 42 days plus additional 30 days.
Arm/Group | Carbamazepine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/35 | 1/35
Other Adverse Events (participants affected / at risk) | 29/35 | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbamazepine (N=35) | Placebo (N=35)
Blood & lymphatic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
General disorders & administration conditions (General disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lab Investigations (Investigations) | 1 (1) | 0 (0)
Nervous system (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbamazepine (N=35) | Placebo (N=35)
Cardiac disprders (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (5) | 2 (2)
General disorders & administration conditions (General disorders) | 3 (3) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lab results (Investigations) | 3 (3) | 0 (0)
Metabolic (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nervous system (Nervous system disorders) | 20 (20) | 11 (11)
Psychiatric (Psychiatric disorders) | 9 (9) | 5 (5)
Skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Vascular (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No